CLINICAL TRIAL: NCT01168024
Title: PRESERV (Prospective Randomized Evaluation to Study the Effects of Reduced Contrast Media on the Vitality of the Kidney) Pivotal Trial
Brief Title: Contrast Media Reduction and Removal in Patients With Chronic Kidney Disease (CKD) (PRESERV)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study closed by sponsor prior to completing enrollment goal.
Sponsor: Osprey Medical, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: TP-6142
Record Dates: First submitted 2010-07-20; First posted 2010-07-22 (Estimated); Results first posted 2016-12-12 (Estimated); Last update posted 2016-12-12 (Estimated); Status verified 2016-10

CONDITIONS: Radiographic Contrast Agent Nephropathy
Keywords: Acute Kidney Injury; Iodinated Contrast Agent Retrieval; Coronary Sinus Cannulation
MeSH Terms: conditions — Acute Kidney Injury | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CINCOR™ System Treatment (Experimental): Use of the CINCOR™ System and CCS-1 device during the pericutanous coronary intervention (PCI) procedure plus Standard of Care peri-procedural hydration for the prevention of contrast induced nephropathy (CIN).
  Interventions: Device: CINCOR™ System and contrast conservation unit (CCS-1); Other: Standard of Care plus peri-procedural hydration
- Standard of Care (Other): The control group will receive a peri and post-procedural hydration rate.
  Interventions: Other: Standard of Care plus peri-procedural hydration

INTERVENTIONS:
Device: CINCOR™ System and contrast conservation unit (CCS-1) — Catheter based system to reduce and remove contrast media and contrast modulator to reduce contrast media
  Arms: CINCOR™ System Treatment
Other: Standard of Care plus peri-procedural hydration — The control group will receive a peri and post-procedural hydration rate.

SUMMARY:
The purpose of this clinical trial is to demonstrate the efficacy and safety of the Osprey Medical CINCOR™ Contrast Removal System.

DETAILED DESCRIPTION:
The CINCOR™ Catheter System to retrieve contrast media from the coronary sinus following injection during percutaneous coronary interventions.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is at least 18 years of age.
2. The subject is a candidate for a therapeutic coronary PCI procedure of the left coronary artery and/or its branches or a combination procedure including left coronary artery/branches AND right coronary artery that is expected to utilize at least 50 mL of iodinated contrast media.
3. The subject has baseline eGFR between 20 and 30 mL/min/1.73 m2 inclusive (as determined by the MDRD equation (Levey 1993)); or patient has eGFR above 30 but less than or equal to 60 with at least two of the following: stage III/IV NYHA congestive heart failure, diabetes mellitus, hypertension, age of at least 75 years.
4. The subject (or subject's legal representative) is willing and able to provide appropriate informed consent.
5. The subject is willing and able to comply with the requirements of the study protocol, including the predefined follow-up evaluations.

Exclusion Criteria:

1. The subject has unstable renal function (acute renal failure or change in serum creatinine of > 0.5mg/dL or > 25% within 7 days of the procedure not attributed to hydration therapy).
2. The subject requires dialysis.
3. The subject has received contrast media within 7 days of the procedure.
4. The subject will receive > 10 ml of iodinated contrast media in any location other than the coronary arteries (e.g. ventriculography, aortography, renal angiography) during the procedure or within a period of 30 days after the procedure.
5. The subject requires one or more of the following nephrotoxic agents: Aminoglycoside antibiotics, Sulfonamides, Amphotericin B, Levofloxacin, Ciprofloxacin, Rifampin, Tetracycline, Intravenous Acyclovir, Pentamidine, Penicillin and Cephalosporins, Cisplatin, Methotrexate, Mitomycin, Cyclosporine, Tacrolimus.
6. The subject has hemoglobin (Hb) < 9.5 g/dL within one (1) week of the procedure.
7. The subject is hemodynamically unstable or requires hemodynamic support including intra-venous inotropes, vasopressors, or any type of ventricular assist devices (including intra-aortic balloon pumps, the Impella cardiac assist device, the TandemHeart VAD, and surgically implanted ventricular assist devices).
8. The subject has had acute myocardial infarction within last 24 hours (as defined in the "Universal Definition of Myocardial Infarction (Thygesen 2007) or has biomarkers of cardiac injury that have not stabilized. (Patients with MI within 96 hours of index procedure must demonstrate falling biomarkers of cardiac injury).
9. The subject has any of the following procedural contra-indications

   1. has a left heart pacing lead or other implant indwelling in the coronary sinus or has had an artificial valve or pacemaker lead implanted in the right heart within 8 weeks of the planned procedure
   2. has a known bleeding diathesis (e.g. thrombocytopenia [<100,000 cells/mm3], heparin-induced thrombocytopenia, hemophilia, or von Willebrand disease, any history of intracranial bleeding, or gastrointestinal or gross genitourinary bleeding)
   3. The subject is currently on intravenous anti-coagulation that cannot be discontinued prior to the procedure
   4. The subject has a known hypersensitivity to both heparin and bivalirudin or aspirin or all thienopyridine agents or iodinated contrast that cannot be adequately pre-medicated
   5. The subject has an active systemic infection
   6. The subject refuses to accept blood products (e.g. Jehovah's Witness)
10. The subject is known to be or suspected to be pregnant, or is lactating (all women of child-bearing potential must have a negative pregnancy test within 72 hours before participating in this protocol).
11. The subject is currently participating in another investigational device or drug study that has not reached its primary endpoint.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2012-12; Primary Completion 2013-10 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregg Stone, MD, Principal Investigator — CRF
Locations (21):
- United States (20):
  - Heart Care Research, LLC, Huntsville, Alabama
  - St. Luke's Medical Center, Phoenix, Arizona
  - Kaiser Permanente, Los Angeles, California
  - Stanford Hospitals and Clinics, Stanford, California
  - Harbor UCLA, Torrance, California
  - The Heart and Vascular Institute of Florida, Clearwater, Florida
  - Infinity Clinical Research, Hollywood, Florida
  - Saint Joseph's Hospital of Atlanta, Atlanta, Georgia
  - Franciscan St. Francis Health, Indianapolis, Indiana
  - St. Mary's Medical Center, Duluth, Minnesota
  - Elyria Memorial Hospital Medical Center, Elyria, Ohio
  - Oklahoma Foundation for Cardiovascular Research, Oklahoma City, Oklahoma
  - York Hospital, York, Pennsylvania
  - South Carolina Heart Center, Columbia, South Carolina
  - Greenville Health System, Greenville, South Carolina
  - Tennova Healthcare - Turkey Creek Medical Center, Knoxville, Tennessee
  - The Methodist Hospital of Research, Houston, Texas
  - Cardiovascular Associates of East Texas, PA, Tyler, Texas
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - Charleston Area Medical Center, Charleston, West Virginia
- Cardiology Center Leipzig Ltd., Leipzig, Saxony, Germany

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- CINCOR™ System and CCS-1: Use of the CINCOR™ System and CCS-1 device during the PCI procedure plus Standard of Care peri-procedural hydration for the prevention of CIN.
- Standard of Care Plus Peri-procedural Hydration: Peri-procedural hydration utilized prior to standard of care PCI.
Period: Overall Study
Arm/Group | CINCOR™ System and CCS-1 | Standard of Care Plus Peri-procedural Hydration
Started | 13 (13 tx/3 controls. Roll-ins occurred for product training, several more treatment cases than control.) | 3
Completed | 13 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Enrollment allowed for both non-randomized roll-in and randomized subjects. Up to three roll-in subjects (maximum of 150 in the trial) were allowed per center to address learning curve issues associated with the coronary sinus cannulation technique and device use.
Groups:
- CINCOR™ System Treatment: Use of the CINCOR™ System and CCS-1 device during the PCI procedure plus Standard of Care peri-procedural hydration for the prevention of CIN.
  CINCOR™ System and CCS-1: Catheter based system to reduce and remove contrast media and contrast modulator to reduce contrast media
  Peri-procedural hydration: The control group will receive a peri and post-procedural hydration rate.
- Standard of Care: Peri-procedural hydration with isotonic saline or sodium bicarbonate for at least 2 hours prior to the procedure and 6-12 hours post-procedure.
  Peri-procedural hydration: The control group will receive a peri and post-procedural hydration rate.
- Total: Total of all reporting groups
Arm/Group | CINCOR™ System Treatment | Standard of Care | Total
Number analyzed (Participants) | 13 | 3 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.2 (11.5) | 82 (13.8) | 71 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 10 | 2 | 12

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Contrast Induced Nephropathy (CIN) in Subjects.
Description: CIN is defined as a post-procedure relative serum creatinine increase ≥ 25% or an absolute serum creatinine increase of ≥ 0.5 mg/dL).
Time Frame: Through 72 hours post-procedure
Measure: Number; unit: participants
Groups:
- Treatment (Roll In and Randomized): CINCOR, CCS-1 and Peri-procedure hydration
- Control: Peri-procedure hydration
Arm/Group | Treatment (Roll In and Randomized) | Control
Number analyzed (Participants) | 13 | 3
participants | 2 | 1

2. Primary Outcome: Evaluating Bleeding/Transfusion Events.
Description: Bleeding/transfusion events evaluated:
  * Blood loss requiring transfusion of ≥ 2 units
  * Thrombolysis in Myocardial Infarction (TIMI) Major Bleeding
  * TIMI Minor Bleeding
Time Frame: Through 30 days post-procedure
Measure: Number; unit: events
Arm/Group | Treatment (Roll In and Randomized) | Control
Number analyzed (Participants) | 13 | 3
events | 0 | 0

3. Primary Outcome: Evaluating Local Events.
Description: Events evaluated include:
  * Coronary sinus perforation, dissection, or occlusion that requires treatment or results in MI or death
  * Pericardial effusions (including pericardial tamponade) requiring treatment
Time Frame: Through 30 days post-procedure.
Measure: Number; unit: events
Arm/Group | Treatment (Roll In and Randomized) | Control
Number analyzed (Participants) | 13 | 3
events | 0 | 0

4. Secondary Outcome: Change in Kidney Function Between the Randomized Groups.
Time Frame: Up to 96 hours post-procedure
Population: Change in eGFR was available for 2 treatment and 1 control subject. 1 out of range eGFR value for a subject (0.1) was not used as this value is not clinically feasible.
Measure: Mean (Standard Deviation); unit: mL/min/1.73m^2
Arm/Group | Treatment (Roll In and Randomized) | Control
Number analyzed (Participants) | 1 | 2
mL/min/1.73m^2 | -6.33 (1.10) | -6.95 (3.61)

ADVERSE EVENTS:
Time Frame: Adverse events were reported through the 30 day follow up period.
Arm/Group | Treatment (Roll In and Randomized) | Control
Serious Adverse Events (participants affected / at risk) | 2/13 | 0/3
Other Adverse Events (participants affected / at risk) | 3/13 | 0/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Roll In and Randomized) (N=13) | Control (N=3)
STEMI (Cardiac disorders) | 1 (1) | 0 (0)
Dizziness (Cardiac disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Roll In and Randomized) (N=13) | Control (N=3)
Chest Pain (Cardiac disorders) | 1 (1) | 0 (0)
Troponin Elevation (Cardiac disorders) | 1 (1) | 0 (0)
Minor Bleeding (Cardiac disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No